CLINICAL TRIAL: NCT01360216
Title: Cluster, Randomized Trial on Provider LARC Education and Training
Brief Title: Cluster, Randomized Trial on Long Acting Reversible Contraception (LARC) Education and Training
Acronym: LARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010-5442
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Contraception Behavior
Keywords: Long-acting reversible contraception; Intrauterine contraception; Intrauterine devices; Single-rod implant; Hormonal contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LARC education and training (Experimental): Clinicians and contraceptive educators practicing in clinics assigned to this arm receive a special half-day Continuing Medical Education (CME/CEU) accredited LARC education and training session.
  Interventions: Behavioral: LARC education and training
- Standard practice- control (No Intervention): Clinicians and contraceptive educators practicing in clinics assigned to this arm do not receive special LARC training and education session. Standard practice will be followed at clinics assigned to the control arm.

INTERVENTIONS:
Behavioral: LARC education and training — A CME/CEU accredited Grand Rounds education and training session will be given to clinicians and contraceptive educators practicing in clinics assigned to the intervention arm. Clinicians will have hands-on training as well. The half-day session emphasizes evidence-based contraceptive counseling and provision.
  Arms: LARC education and training

SUMMARY:
The purpose of the study is to measure whether an education and training intervention for clinicians and contraceptive counselors on long-acting reversible contraception (LARC) will result in greater use of the methods among contraceptive patients.

DETAILED DESCRIPTION:
Unintended pregnancy is extremely high in the United States among young women, and use of contraceptives with top-tier effectiveness, intrauterine contraception and implants, is low. Contraceptive providers in the US have low knowledge of current scientific evidence on LARC methods, and do not routinely include these methods in counseling patients at highest risk of unintended pregnancy. This intervention provides evidence-based education and hands-on training to clinicians and contraceptive educators in Planned Parenthood affiliated Title X clinics throughout the US on LARC methods.

ELIGIBILITY:
Inclusion Criteria:

This study involves two groups of human subjects: patients and staff at participating Planned Parenthood (PP) clinics in the United States.

Patient participants are young women receiving contraceptive counseling at Planned Parenthood clinics and staff participants are the clinicians and health educators serving these women.

Patients must be:

Female;

* Age 18-25;
* Fluent in English or Spanish;
* Not wanting to become pregnant in the next 12 months;
* Sexually active in past 3 months;
* At risk of pregnancy;
* Received contraceptive counseling;
* Not pregnant;
* Willing to be contacted by telephone over the next 12 months.

Clinic staff must be:

* Employed by a participating PP clinic; and
* Offer clinical care, counseling or education for abortion or contraception at the clinic. (This may include physicians, advance practice clinicians, nurses, social workers and health educators.)

For clinics to be eligible to be study sites, they must:

* Not share staff
* Have no active LARC interventions ongoing
* Have >400 clients/year

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of contraceptive patients choosing a LARC method | Baseline
  We are measuring the proportion of patients deciding to use a LARC method at intervention and control clinics in a patient cohort aged 18-25 years (n=1500). We are also measuring with clinic service statistics the proportion of contraceptive patients selecting LARC v. non-LARC methods during the 12 month-period before the intervention and the 12-month period after the intervention, to supplement the analysis with individual patient data.

SECONDARY OUTCOMES:
Unintended pregnancy | 12 months
  We are measuring unintended pregnancy among contraceptive patients receiving contraceptive counseling at intervention and control clinics (total number 1,500) during a 12 month period.

OTHER OUTCOMES:
Sub-analysis for primary outcome, decision to use LARC method | Baseline
  We will assess the outcome decision to use LARC, by important factors affecting contraceptive methods, including policy variables for contraceptive coverage (Medicaid expansion waiver states, mandates for contraceptive coverage for private insurance), clinic visit type (post-abortion or family planning), pregnancy intentions, mental health and domestic violence, male partner, provider-patient interaction, sociodemographic factors (age, race/ethnicity, education).
Sub-analyses for pregnancy during 12-month study | 12 months (Baseline to 12-month Follow-up)
  We will assess the secondary outcome, pregnancy during 12-month study, by important pregnancy risk variables, including clinic visit type (post-abortion or family planning), pregnancy intentions, mental health and domestic violence, provider-patient interaction, male partner, sociodemographic (age, race/ethnicity, education) and policy variables (Medicaid expansion waiver states, mandates for contraceptive coverage for private insurance).
Provider LARC knowledge and practices | Baseline and 12-month Follow-up
  We will measure providers' LARC knowledge and practices (discuss LARC methods with contraceptive clients) at baseline and 12-month follow-up, using provider survey data) to assess whether they integrate LARC into standard clinic practice in the intervention arm.
LARC use over time | 12 months (baseline to 12 month follow-up)
  We will measure patient use of LARC methods with patient data (n=1500) over the course of the study, and assess factors associated with continued use over time, including sociodemographic, reproductive, mental health, and contraceptive policy factors.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia C Harper, PhD, Principal Investigator — University of California San Francisco School of Medicine; J. Joseph Speidel, MD, MPH, Principal Investigator — University of California San Francisco School of Medicine
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Thompson KM, Speidel JJ, Saporta V, Waxman NJ, Harper CC. Contraceptive policies affect post-abortion provision of long-acting reversible contraception. Contraception. 2011 Jan;83(1):41-7. doi: 10.1016/j.contraception.2010.06.008. Epub 2010 Sep 20. PMID 21134502
- [Background] Harper CC, Blum M, de Bocanegra HT, Darney PD, Speidel JJ, Policar M, Drey EA. Challenges in translating evidence to practice: the provision of intrauterine contraception. Obstet Gynecol. 2008 Jun;111(6):1359-69. doi: 10.1097/AOG.0b013e318173fd83. PMID 18515520
- [Background] Speidel JJ, Harper CC, Shields WC. The potential of long-acting reversible contraception to decrease unintended pregnancy. Contraception. 2008 Sep;78(3):197-200. doi: 10.1016/j.contraception.2008.06.001. Epub 2008 Jul 9. No abstract available. PMID 18692608
- [Background] Goodman S, Hendlish SK, Reeves MF, Foster-Rosales A. Impact of immediate postabortal insertion of intrauterine contraception on repeat abortion. Contraception. 2008 Aug;78(2):143-8. doi: 10.1016/j.contraception.2008.03.003. Epub 2008 May 14. PMID 18672116
- [Background] Goodman S, Hendlish SK, Benedict C, Reeves MF, Pera-Floyd M, Foster-Rosales A. Increasing intrauterine contraception use by reducing barriers to post-abortal and interval insertion. Contraception. 2008 Aug;78(2):136-42. doi: 10.1016/j.contraception.2008.03.008. Epub 2008 Jun 18. PMID 18672115
- [Background] Kavanaugh ML, Jones RK, Finer LB. How commonly do US abortion clinics offer contraceptive services? Contraception. 2010 Oct;82(4):331-6. doi: 10.1016/j.contraception.2010.04.010. Epub 2010 May 21. PMID 20851226
- [Background] Kavanaugh ML, Jones RK, Finer LB. Perceived and insurance-related barriers to the provision of contraceptive services in U.S. abortion care settings. Womens Health Issues. 2011 May-Jun;21(3 Suppl):S26-31. doi: 10.1016/j.whi.2011.01.009. PMID 21530835
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Hladky KJ, Allsworth JE, Madden T, Secura GM, Peipert JF. Women's knowledge about intrauterine contraception. Obstet Gynecol. 2011 Jan;117(1):48-54. doi: 10.1097/AOG.0b013e318202b4c9. PMID 21173643
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] Madden T, Allsworth JE, Hladky KJ, Secura GM, Peipert JF. Intrauterine contraception in Saint Louis: a survey of obstetrician and gynecologists' knowledge and attitudes. Contraception. 2010 Feb;81(2):112-6. doi: 10.1016/j.contraception.2009.08.002. Epub 2009 Sep 16. PMID 20103447
- [Background] Kittur ND, Secura GM, Peipert JF, Madden T, Finer LB, Allsworth JE. Comparison of contraceptive use between the Contraceptive CHOICE Project and state and national data. Contraception. 2011 May;83(5):479-85. doi: 10.1016/j.contraception.2010.10.001. Epub 2010 Nov 23. PMID 21477693
- [Background] Fleming KL, Sokoloff A, Raine TR. Attitudes and beliefs about the intrauterine device among teenagers and young women. Contraception. 2010 Aug;82(2):178-82. doi: 10.1016/j.contraception.2010.02.020. Epub 2010 Apr 13. PMID 20654760
- [Background] Darney P, Patel A, Rosen K, Shapiro LS, Kaunitz AM. Safety and efficacy of a single-rod etonogestrel implant (Implanon): results from 11 international clinical trials. Fertil Steril. 2009 May;91(5):1646-53. doi: 10.1016/j.fertnstert.2008.02.140. Epub 2008 Apr 18. PMID 18423453
- [Background] Raine TR, Foster-Rosales A, Upadhyay UD, Boyer CB, Brown BA, Sokoloff A, Harper CC. One-year contraceptive continuation and pregnancy in adolescent girls and women initiating hormonal contraceptives. Obstet Gynecol. 2011 Feb;117(2 Pt 1):363-371. doi: 10.1097/AOG.0b013e31820563d3. PMID 21252751
- [Background] Shelton JD. Risk of clinical pelvic inflammatory disease attributable to an intrauterine device. Lancet. 2001 Feb 10;357(9254):443. doi: 10.1016/S0140-6736(00)04012-5. PMID 11273068
- [Background] Grimes DA, Lopez LM, Schulz KF, Stanwood NL. Immediate postabortal insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD001777. doi: 10.1002/14651858.CD001777.pub3. PMID 20556754
- [Background] Allen RH, Goldberg AB, Grimes DA. Expanding access to intrauterine contraception. Am J Obstet Gynecol. 2009 Nov;201(5):456.e1-5. doi: 10.1016/j.ajog.2009.04.027. Epub 2009 Jun 13. PMID 19527902
- [Background] Deans EI, Grimes DA. Intrauterine devices for adolescents: a systematic review. Contraception. 2009 Jun;79(6):418-23. doi: 10.1016/j.contraception.2008.12.009. Epub 2009 Feb 7. PMID 19442775
- [Background] Grimes DA. Intrauterine device and upper-genital-tract infection. Lancet. 2000 Sep 16;356(9234):1013-9. doi: 10.1016/S0140-6736(00)02699-4. PMID 11041414
- [Background] Stanwood NL, Garrett JM, Konrad TR. Obstetrician-gynecologists and the intrauterine device: a survey of attitudes and practice. Obstet Gynecol. 2002 Feb;99(2):275-80. doi: 10.1016/s0029-7844(01)01726-4. PMID 11814509
- [Background] Postlethwaite D, Shaber R, Mancuso V, Flores J, Armstrong MA. Intrauterine contraception: evaluation of clinician practice patterns in Kaiser Permanente Northern California. Contraception. 2007 Mar;75(3):177-84. doi: 10.1016/j.contraception.2006.10.010. Epub 2007 Jan 16. PMID 17303486
- [Background] Hubacher D, Vilchez R, Gmach R, Jarquin C, Medrano J, Gadea A, Grey T, Pierre-Louis B. The impact of clinician education on IUD uptake, knowledge and attitudes: results of a randomized trial. Contraception. 2006 Jun;73(6):628-33. doi: 10.1016/j.contraception.2006.02.003. Epub 2006 Mar 29. PMID 16730497
- [Background] Hubacher D, Lara-Ricalde R, Taylor DJ, Guerra-Infante F, Guzman-Rodriguez R. Use of copper intrauterine devices and the risk of tubal infertility among nulligravid women. N Engl J Med. 2001 Aug 23;345(8):561-7. doi: 10.1056/NEJMoa010438. PMID 11529209
- [Background] Trussell J, Lalla AM, Doan QV, Reyes E, Pinto L, Gricar J. Cost effectiveness of contraceptives in the United States. Contraception. 2009 Jan;79(1):5-14. doi: 10.1016/j.contraception.2008.08.003. Epub 2008 Sep 25. PMID 19041435
- [Derived] Steinberg JR, Adler NE, Thompson KM, Westhoff C, Harper CC. Current and past depressive symptoms and contraceptive effectiveness level method selected among women seeking reproductive health services. Soc Sci Med. 2018 Oct;214:20-25. doi: 10.1016/j.socscimed.2018.08.009. Epub 2018 Aug 13. PMID 30138841
- [Derived] Rocca CH, Goodman S, Grossman D, Cadwallader K, Thompson KMJ, Talmont E, Speidel JJ, Harper CC. Contraception after medication abortion in the United States: results from a cluster randomized trial. Am J Obstet Gynecol. 2018 Jan;218(1):107.e1-107.e8. doi: 10.1016/j.ajog.2017.09.020. Epub 2017 Oct 3. PMID 28986072
- [Derived] Gibbs SE, Rocca CH, Bednarek P, Thompson KMJ, Darney PD, Harper CC. Long-Acting Reversible Contraception Counseling and Use for Older Adolescents and Nulliparous Women. J Adolesc Health. 2016 Dec;59(6):703-709. doi: 10.1016/j.jadohealth.2016.07.018. Epub 2016 Sep 21. PMID 27665153